CLINICAL TRIAL: NCT00749840
Title: Attitudes and Beliefs and the Steps of HIV Care
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2008-0011
Record Dates: First submitted 2008-09-05; First posted 2008-09-09 (Estimated); Last update posted 2013-02-13 (Estimated); Status verified 2013-02

CONDITIONS: Human Immunodeficiency Virus Infections
Keywords: Acquired Immune Deficiency Syndrome; Human Immunodeficiency Virus; Questionnaire; AIDS; HIV; Highly Active Antiretroviral Therapy; HAART; Steps of HIV Care; CDC
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HIV Care Questionnaire: Patients with a new diagnosis of HIV infection.
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — Questionnaire taking 60-90 minutes.
  Other Names: Survey

SUMMARY:
Through a prospective observational cohort study enrolling patients newly diagnosed with Human immunodeficiency virus (HIV):

Aim 1: Assess attitudes and beliefs about HIV disease and care over time and relate those attitudes and beliefs to success in following the Steps of HIV Care.

Aim 2: Validate a simple visual analogue scale for assessing adherence to highly active antiretroviral therapy (HAART) in patients newly starting HAART in routine care.

Aim 3: Implement latent growth curve analysis for modeling changes in attitudes and beliefs over time, and for assessing the impact of the components of the Steps of HIV Care model on health outcomes.

DETAILED DESCRIPTION:
The introduction of highly active antiretroviral therapy (HAART) dramatically improved the survival of patients with HIV in the US. The effectiveness of HAART in routine care is determined by the success with which patients are able to follow certain crucial Steps of HIV Care. This 'Steps of HIV Care' framework is based on the Centers for Disease Control and Prevention's (CDC's) "Serostatus Approach to Fighting the HIV Epidemic," which has been overlaid with patient and process of care factors. It includes 1) access outpatient care, 2) utilize care and treatment services, and 3) adhere to care, including medications and appointments.

ELIGIBILITY:
Inclusion Criteria:

* A new diagnosis of HIV infection, defined as diagnosed with HIV less than 3 months before the current diagnosis AND not yet having completed a regularly scheduled outpatient primary medical care visit for HIV.
* Ability to speak English or Spanish. Ability to provide informed consent (or have a representative able to do so). Age greater than or equal to 18 years.
* Adherence Sub-Study. Persons in the Steps of HIV Care Cohort Study and prescribed HAART at either Thomas Street Health Center, the Northwest Health Center, or the Michael E. DeBakey VA HIV Clinic. Using or planning on using the Thomas Street Health Center, Northwest Health Center or the Michael E. DeBakey VA pharmacy to fill their prescriptions for HAART. On HAART for less than 6 months at the time of enrollment into the sub-study.
* Qualitative Sub-Study Persons in Steps of HIV Care Cohort. Willing and cognitively able to complete the interview, in the eyes of the investigator or the research team.

Exclusion Criteria:

* Persons diagnosed with HIV more than 3 months before the current diagnosis will be excluded, as will persons diagnosed with HIV less than 3 months before the current diagnosis who have seen an outpatient provider for HIV care at a regularly scheduled visit.
* Patients with dementia, active psychosis, or other conditions that will not allow them to accurately complete the interview will be followed separately from the main cohort, provided informed consent can be obtained from their representative.
* Since the instruments are interviewer-administered, illiterate patients will not be excluded; in that circumstance, the research staff will read the informed consent documents to the potential participant.
* Patients who speak neither English nor Spanish will be excluded, since the informed consent and survey instruments will be available in only those languages. Pregnant women will not be excluded, as the study poses no risk to the fetus.
* Adherence Sub-Study. As for the Steps of HIV Care Cohort Study. In addition: Patients will be excluded if they are not willing to forego use of a pill organizer for the medication to be monitored with the computerized caps. Pill organizers for the unmonitored medications will be allowed. Patients will be excluded if they are not themselves responsible for taking their own medication, i.e., if they are institutionalized or incarcerated (though neither Thomas Street Health Center, Northwest Health Center, nor the VA HIV Clinic cares for incarcerated person).
* Or, if a person other than the patient takes primary responsibility for ensuring medication is taken by the patient. We will also exclude patients who cannot agree to not pocket doses on a routine basis, that is, remove extra pills from the bottle for later ingestion. This behavior will likely be infrequently practiced, since almost all HAART regimens currently are once or twice daily rather than thrice daily.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a new diagnosis of HIV infection.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-04; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Survey to Assess Attitudes + Beliefs about Steps of HIV Disease Care | Interviewer-administered at time of enrollment and every 3 months for 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Kallen, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org